CLINICAL TRIAL: NCT03460145
Title: Lavender Aromatherapy; Its Effect on Preoperative Anxiety and Propofol Requirement for Anaesthesia.
Brief Title: Lavender Oil on Preoperative Anxiety and Sedation Requirement in General Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 37839
Record Dates: First submitted 2018-01-24; First posted 2018-03-09 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2018-04

CONDITIONS: Preoperative Anxiety
Keywords: Lavender Oil,; Propofol
MeSH Terms: interventions — lavender oil; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strip with Lavender Oil (Lx) (Experimental): Application of Nasal Strip with essential oil (Lavender), 20minutes before induction.
  VAS- Anxiety scores pre and post inhalation.
  Interventions: Other: Lavender Oil on Nasal Strip (Lx); Drug: Propofol 1 % Injectable Suspension
- Strip without Lavender Oil (Px) (Placebo Comparator): Application of Nasal strip without essential oil, acting as placebo. VAS- Anxiety scores pre and post placebo.
  Interventions: Other: Strip without Lavender Oil (Px); Drug: Propofol 1 % Injectable Suspension

INTERVENTIONS:
Other: Lavender Oil on Nasal Strip (Lx) — Usage of Aromatherapy for Preoperative Anxiety
  Arms: Strip with Lavender Oil (Lx)
Other: Strip without Lavender Oil (Px) — Strip without Lavender Oil (Px)
  Arms: Strip without Lavender Oil (Px)
Drug: Propofol 1 % Injectable Suspension — Propofol 1% (10mg/mL)

SUMMARY:
Assessment of how Lavender oil reduces preoperative anxiety and subsequently influences requirement of induction agents for general anesthesia.

DETAILED DESCRIPTION:
This study aims to use aromatherapy (Lavender oil) to reduce Preoperative Anxiety among Female patients coming for elective surgeries under General Anesthesia.

As a consequence of that, the effect is also evaluated on how that influences the amount of intravenous sedation is required during induction for General Anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Female

Exclusion Criteria:

* Patients on B-blockers and or antidepressants.
* BMI > 35kg/m2
* History of atopy
* History of alcoholism, substance abuse, smoking
* Patients with cancer

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — For General Surgery
Enrollment: 108 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
1. Visual Analog Scoring for Anxiety | 1 day
  Self reported anxiety score before and after inhalation of aromatherapy. 3 questions about preoperative anxiety are asked and scoring is done based on a 0-10cm scale (0= no anxiety, 10= agonizing anxiety). Cumulative scores for all 3 questions above 5 indicates preoperative anxiety.

SECONDARY OUTCOMES:
1. Amount of sedation used to achieve Loss of Consciousness | Less than 30minutes
  Induction for general anesthesia using Target control Infusion of Propofol 1% (10mg/mL) using the Schnider protocol, administered via a TIVA Agilia infusion pump to achieve a target plasma concentration of 4mcg/ml until loss of consciousness.

CONTACTS AND LOCATIONS:
Overall Officials: Raha Abdul Rahman, MD, Principal Investigator — Consultant Anesthesiologist
Locations (1):
- University Kebangsaan Malaysia, Kuala Lumpur, Cheras, Malaysia

IPD SHARING:
Plan to Share IPD: No